CLINICAL TRIAL: NCT00605527
Title: Targeted Genomic Analysis of Coagulation Pathways in Acute Lung Injury
Brief Title: Understanding the Role of Genes and Biomarkers in the Inflammation and Blood Clotting Process in Children With Acute Lung Injury
Acronym: PALI
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 545; K23HL085526 (NIH); K23HL085526-01A1 (NIH)
Record Dates: First submitted 2008-01-18; First posted 2008-01-31 (Estimated); Last update posted 2020-07-20 (Actual); Status verified 2020-07

CONDITIONS: Respiratory Distress Syndrome, Adult
Keywords: Acute Lung Injury; Acute Respiratory Distress Syndrome
MeSH Terms: conditions — Respiratory Distress Syndrome; Acute Lung Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and plasma samples will be analyzed
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Acute lung injury (ALI)/Acute Respiratory Distress Syndrome (ARDS) is a severe lung condition that causes respiratory failure. This study will examine if differences in genes and biomarkers involved in the inflammation and blood clotting process may affect the severity of and recovery from ALI/ARDS in children hospitalized with the condition.

DETAILED DESCRIPTION:
ALI/ARDS is a life-threatening condition that involves inflammation of the lungs and fluid accumulation in the air sacs, which leads to low blood oxygen levels and respiratory failure. Common causes include pneumonia, sepsis, and lung trauma. Symptoms, including breathing difficulty, low blood pressure, and organ failure, usually develop within 24 to 48 hours of the original injury or illness. Most patients require immediate care in an intensive care unit, and the main form of treatment is mechanical ventilation, which delivers oxygen and a continuous level of pressure to the damaged lungs. Although progress has been made in understanding how ALI/ARDS develops, it is still unknown why recovery outcomes differ among people. Differences in the genetic basis of protein C and fibrinolysis pathways, which both play a role in preventing blood clots, may be a factor in determining the severity of and recovery from ALI. The purpose of this study is to analyze plasma and DNA from children with ALI/ARDS to identify biomarkers and genetic variations that may be related to clinical outcomes.

This study will enroll children who are hospitalized with ALI/ARDS. Participants' medical records will be reviewed to gather information about symptoms, physical exam findings, mechanical ventilator settings, and laboratory test results. A blood collection will occur on Days 1 and 3. Study researchers will analyze plasma biomarkers and use high throughput DNA sequencing technology to analyze participants' DNA.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized and requiring supplemental oxygen
* Meets the American-European consensus definition of ALI/ARDS, defined as partial pressure of oxygen in arterial blood/fraction of inspired oxygen (PaO2/FiO2) ratio of less than 300 mm Hg, bilateral opacities on a chest radiograph, and either a pulmonary wedge pressure of less than 18 mm Hg or the absence of clinical evidence of left atrial hypertension
* Acute pulmonary parenchymal disease (i.e., onset of bilateral infiltrates on chest radiograph within 48 hours of screening)
* PaO2/FiO2 less than or equal to 300 mm Hg, regardless of the mean airway pressure
* At least one arterial blood gas confirming partial pressure of oxygen/fraction of inspired oxygen (PO2/FiO2) ratio less than 300 mm Hg or Fi02/Sao2 on pulse oximetry of less than 320

Exclusion Criteria:

* Clinical signs of left ventricular failure, pulmonary capillary wedge pressure greater than 18 mm Hg, or evidence, such as echocardiography, suggesting a cardiac basis for the pulmonary edema
* Presence of right-to-left intracardiac shunt

Ages: 30 Days to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients who are admitted to the University of California, San Francisco hospital and participating sites including Children's Hospital of Oakland with ALI/ARDS.
Sampling Method: Non-Probability Sample
Enrollment: 396 (Actual)
Dates: Start 2007-11; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Number of ventilator-free days | Measured during participant's hospital stay

SECONDARY OUTCOMES:
Mortality and organ dysfunction | Measured during participant's hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Anil Sapru, MD, MAS, Principal Investigator — University of California, San Francisco
Locations (5):
- United States (5):
  - Children's Hospital Central California, Fresno, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Children's Hospital & Research Center of Oakland, Oakland, California
  - University of California, San Francisco, San Francisco, California
  - American Family Children's Hospital, Madison, Wisconsin